CLINICAL TRIAL: NCT01171924
Title: A Phase Ib Open Label, Expansion Study to Investigate the Safety, Efficacy, and Pharmacokinetics of Intravenous CUDC-101 in Subjects With Advanced Head and Neck, Gastric, Breast, Liver and Non-small Cell Lung Cancer Tumors
Brief Title: A Phase Ib Expansion Study Investigating the Safety, Efficacy, and Pharmacokinetics of Intravenous CUDC-101 in Subjects With Advanced Head and Neck, Gastric, Breast, Liver and Non-small Cell Lung Cancer Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUDC-101-102
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Head and Neck Cancer; Liver Cancer; Breast Cancer; Gastric Cancer; Non-Small Cell Lung Cancer
Keywords: Head and Neck Cancer; Liver Cancer; Breast Cancer; Gastric Cancer; Non-Small Cell Lung Cancer; EGFR; HDAC; Her2; CUDC-101
MeSH Terms: conditions — Head and Neck Neoplasms; Liver Neoplasms; Breast Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — 7-(4-(3-ethynylphenylamino)-7-methoxyquinazolin-6-yloxy)-N-hydroxyheptanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: 5 days/week schedule (Experimental)
  Interventions: Drug: CUDC-101
- Arm B: 3 days/week schedule (Experimental)
  Interventions: Drug: CUDC-101

INTERVENTIONS:
Drug: CUDC-101 — CUDC-101 administered as a 1 hour intravenous infusion at the maximum tolerated dose of 275 mg/m2 consecutively for 5 days on each 14 day cycle.
  Arms: Arm A: 5 days/week schedule
Drug: CUDC-101 — CUDC-101 administered as a 1 hour intravenous infusion at the maximum tolerated dose of 275 mg/m2 on Monday, Wednesday, Friday for three consecutive weeks of each 28 day cycle.
  Arms: Arm B: 3 days/week schedule

SUMMARY:
This is a phase Ib open label, expansion study of CUDC-101 in patients with advanced head and neck, gastric, breast, liver, and non-small cell lung cancer tumors. CUDC-101 is a multi-targeted agent designed to inhibit epidermal growth factor receptor (EGFR), human epidermal growth factor receptor Type 2 (Her2) and histone deacetylase (HDAC). The study is designed to compare the safety and tolerability of CUDC-101 when administered at the maximum tolerated dose on either a 5 days/week schedule or a 3 days/week schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathologically confirmed diagnosis of advanced breast, gastric, head and neck, liver and non-small cell lung cancer.

  * For subjects with non-small cell lung cancer only:

    * Most recent treatment must be erlotinib and subjects must have had a radiographic partial or complete response to treatment as defined by RECIST criteria and should be currently progressing after the documented response.
    * A documented mutation in EGFR exons 19 or 21
* Subjects must have no further standard of care options or have refused standard therapy
* Measurable or evaluable disease
* Age ≥ 18 years
* ECOG performance < 2
* Life expectancy ≥ 3 months
* If female, neither pregnant or lactating
* If of child bearing potential, must use adequate birth control
* Absolute neutrophil count ≥ 1,500/µL; platelets ≥ 100,000/µL;
* Creatinine ≤ 1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60mL/min/1.73m2
* Total bilirubin ≤ 1.5x ULN; AST/ALT ≤ 2.5x ULN. In subjects with documented liver metastases, the AST/ALT may be ≤ 5x ULN
* Prothrombin time ≤1.5x ULN, unless receiving therapeutic anticoagulation
* Serum magnesium and potassium within normal limits (may use supplements to achieve normal values)
* Subjects with brain metastases are eligible if controlled on a stable dose ≤ 10mg prednisone/day or its equivalent dose of steroids
* Able to render informed consent and to follow protocol requirements.

Exclusion Criteria:

* Anticancer therapy within 4 weeks of study entry.
* Use of investigational agent(s) within 30 days of study entry
* History of cardiac disease with a New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF), myocardial infarction (MI) or unstable angina in the past 6 months prior to Day 1 of treatment, serious arrhythmias requiring medication for treatment.
* Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C. Subjects with liver cancer and hepatitis may be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - San Diego Pacific Oncology and Hematology Associates, Encinitas, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Mountain Blue Global Cancer Care, Wheat Ridge, Colorado
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Lai CJ, Bao R, Tao X, Wang J, Atoyan R, Qu H, Wang DG, Yin L, Samson M, Forrester J, Zifcak B, Xu GX, DellaRocca S, Zhai HX, Cai X, Munger WE, Keegan M, Pepicelli CV, Qian C. CUDC-101, a multitargeted inhibitor of histone deacetylase, epidermal growth factor receptor, and human epidermal growth factor receptor 2, exerts potent anticancer activity. Cancer Res. 2010 May 1;70(9):3647-56. doi: 10.1158/0008-5472.CAN-09-3360. Epub 2010 Apr 13. PMID 20388807
- See also: Curis, Inc. Company Website — http://www.curis.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: 5 Days/Week Schedule | Arm B: 3 Days/Week Schedule
Started | 23 | 23
Completed | 0 | 0
Not Completed | 23 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 5 Days/Week Schedule | Arm B: 3 Days/Week Schedule | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Median (Full Range); unit: years] | 61.0 [40.0 to 78.0] | 65.0 [37.0 to 85.0] | 63.0 [37.0 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 18 | 13 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety and tolerability will be assessed in the two treatment arms and the incidence of adverse events will be compared.
Time Frame: 12-15 months
Measure: Number; unit: participants
Arm/Group | Arm A: 5 Days/Week Schedule | Arm B: 3 Days/Week Schedule
Number analyzed (Participants) | 23 | 23
participants | 23 | 23

ADVERSE EVENTS:
Arm/Group | Arm A: 5 Days/Week | Arm B: 3 Days/Week
Serious Adverse Events (participants affected / at risk) | 12/23 | 9/23
Other Adverse Events (participants affected / at risk) | 23/23 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 5 Days/Week (N=23) | Arm B: 3 Days/Week (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Supraventricular tacycardia (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 5 | 3
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 5 Days/Week (N=23) | Arm B: 3 Days/Week (N=23)
Nausea (General disorders) | 3 | 9
Fatigue (General disorders) | 2 | 7
Vomiting (Gastrointestinal disorders) | 2 | 6
Blood Creatinine Increased (Blood and lymphatic system disorders) | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Decreased Appetite (General disorders) | 4 | 2
Asthenia (General disorders) | 2 | 3
Infusion site phlebitis (Skin and subcutaneous tissue disorders) | 2 | 3
ALP Increased (Blood and lymphatic system disorders) | 0 | 4
ALT Increased (Blood and lymphatic system disorders) | 0 | 4
AST Increased (Blood and lymphatic system disorders) | 0 | 4
BUN Increased (Blood and lymphatic system disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1
Pyrexia (General disorders) | 4 | 0
Hypokalaemia (Blood and lymphatic system disorders) | 2 | 1
Hypomagnesaemia (Blood and lymphatic system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No